CLINICAL TRIAL: NCT00895752
Title: Riluzole in Fragile X Syndrome: A Pilot Study Incorporating Biomarker Assay
Brief Title: Riluzole in Fragile X Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0809-11
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Riluzole (Experimental): Six week open-label treatment with riluzole, maximum dose of 50 mg twice a day.
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Riluzole — Six week open-label treatment with riluzole, maximum dose of 50 mg twice a day.

SUMMARY:
The purpose of this study is to investigate the effectiveness and tolerability of riluzole in adults with Fragile X Syndrome.

DETAILED DESCRIPTION:
Fragile X Syndrome (FXS) represents the most common inherited form of intellectual disability. FXS is more common in males and the symptoms associated with the disorder are more marked in males. FXS is associated with characteristic physical features, behaviors, and comorbidities. Those with FXS often suffer from behavioral difficulties that include anxiety-related symptoms (shyness, social phobia, obsessive-compulsive disorder (OCD) symptoms), attention deficit hyperactivity symptoms (overarousal, hyperactivity, distractibility, impulsivity) and aggressive/self-injurious behaviors.

Riluzole is approved by the FDA for use in treating amyotrophic lateral sclerosis (ALS) in adults. Recently, riluzole has been the subject of several open-label studies describing the use of the drug in treatment-resistant depression and OCD.

Given the overlap between repetitive behavior in FXS and symptoms of OCD, it is logical to study riluzole in FXS given the compound's promise in ameliorating treatment-refractory symptoms of OCD.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 years or older.
* Confirmed molecular diagnosis of Fragile X Syndrome.
* Clinical Global Impression Severity (CGI-S) score of 3 or greater.
* Significant interfering repetitive behavior as determined by the principal investigator.
* Must be in good health as determined by screening procedures including a detailed medical history, and complete physical and neurological examination.
* Dosing of concomitant medications during the study must remain stable.

Exclusion Criteria:

* Pregnancy.
* Concomitant use of another glutamatergic agent (memantine, topiramate, amantadine, among others.
* Evidence of prior trial of riluzole and/or hypersensitivity/allergic reaction to riluzole.
* Abnormal baseline liver function tests at screen or by history; or complete blood count abnormalities at screen or by history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Erickson, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Child and Adolescent Psychiatry Clinic - Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Erickson CA, Weng N, Weiler IJ, Greenough WT, Stigler KA, Wink LK, McDougle CJ. Open-label riluzole in fragile X syndrome. Brain Res. 2011 Mar 22;1380:264-70. doi: 10.1016/j.brainres.2010.10.108. Epub 2010 Nov 5. PMID 21059347

RESULTS

PARTICIPANT FLOW:
Groups:
- Riluzole: 6 subjects received open label riluzole, maximum dose of 50mg bid.
Period: Overall Study
Arm/Group | Riluzole
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Riluzole: Six subjects received 6-weeks of open-label riluzole with maximum dose of 50mg bid.
Arm/Group | Riluzole
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 22.5 [19 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6
Aberrant Behavior Checklist [Mean (Standard Deviation); unit: units on a scale] — The Aberrant Behavior Checklist (ABC) is a 58-item measure of maladaptive behaviors and is used as a measure of drug effects. The ABC has 5 subscales: Social Withdrawal (16 items) ranging from 0 (not at all) to 48 (severe), Irritability (15 items) ranging from 0 (not at all) to 45 (severe), Inappropriate Speech (4 items) ranging from 0 (not at all) to 12 (severe), Hyperactivity (16 items) ranging from 0 (not at all) to 48 (severe), and Stereotypy (7 items) ranging from 0 (not at all) to 21 (severe). Items are rated from 0 (not at all) to 3 (severe).
  units on a scale
    ABC Irritability | 15.2 (11.4)
    ABC Social Withdrawal | 15.8 (11.0)
    ABC Stereotypy | 8.3 (7.8)
    ABC Hyperactivity | 19.5 (8.3)
    ABC Inappropriate Speech | 8.5 (2.7)
ADHD rating scale [Mean (Standard Deviation); unit: units on a scale] — The ADHD Rating Scale is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder. The ADHD Rating Scale-IV is completed by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. The total score can range from 0 to 54, with a higher score indicating greater severity.
  units on a scale | 24.3 (8.4)
Clinical Global Improvement-Severity [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  units on a scale | 4.3 (0.5)
Peabody Picture Vocabulary Test [Mean (Standard Deviation); unit: units on a scale] — The Peabody Picture Vocabulary Test is one of the most commonly used assessment tests that measure verbal ability in standard American English vocabulary. This test has been nationally standardized using examinees from various age groups, from children to adults. Thus, the raw scores are equated to mental age, using the norms obtained from standardization. The total standard scores range from 40 (worse receptive vocabulary) to 160 (better receptive vocabulary). The scores can also be converted to percentile rank.
  units on a scale | 116.8 (40.2)
Social Reciprocity Scale [Mean (Standard Deviation); unit: units on a scale] — The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows: 0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment
  units on a scale | 114.7 (23.6)
Children's Yale-Brown Obsessive Compulsive Scale modified for pervasive developmental disorders [Mean (Standard Deviation); unit: units on a scale] — The Children's Yale-Brown Obsessive Compulsive Scales-Modified (CY-BOCS) is a 5-item, semi-structured clinician rating scale modified designed to rate the current severity of repetitive behavior in children and adolescents with PDD. Once the current repetitive behaviors are identified, they are separately rated on 5 items: Time Spent, Interference, Distress, Resistance, and Control. Each of these items is scored on a 5-point scale form 0 (least symptomatic) to 4 (most symptomatic). The CY-BOCS yields a Total Score from 0 to 20 and is sensitive to change.
  units on a scale | 11.2 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse
Time Frame: Obtained at Week 6
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 6
units on a scale | 3.5 [2 to 4]

2. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Description: The CY-BOCS PDD has been utilized in a largescale clinical treatment study of repetitive behavior in idiopathic ASDs. CYBOCS-PDD scores range from 0 to 20 and measure repetitive/compulsive behavior and not obsessions. Higher score indicate worse outcome.
Time Frame: Obtained at Baseline and Week 6
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Riluzole
Number analyzed (Participants) | 6
Units on a Scale
  Baseline | 11.2 (3.2)
  Six Weeks | 9.7 (3.3)

3. Secondary Outcome: Aberrant Behavior Checklist
Description: The Aberrant Behavior Checklist (ABC) is a 58-item measure of maladaptive behaviors and is used as a measure of drug effects. The ABC has 5 subscales: Social Withdrawal (16 items) ranging from 0 (not at all) to 48 (severe), Irritability (15 items) ranging from 0 (not at all) to 45 (severe), Inappropriate Speech (4 items) ranging from 0 (not at all) to 12 (severe), Hyperactivity (16 items) ranging from 0 (not at all) to 48 (severe), and Stereotypy (7 items) ranging from 0 (not at all) to 21 (severe). Items are rated from 0 (not at all) to 3 (severe).
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 6
units on a scale
  Irritablity | 8.3 (7.7)
  Social Withdrawal | 9.7 (8.0)
  Stereotypy | 5.3 (6.4)
  Hyperactivity | 15.0 (9.2)
  Inappropriate Speech | 6.2 (4.0)

4. Secondary Outcome: The ADHD Rating Scale
Description: The ADHD Rating Scale is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder. The ADHD Rating Scale-IV is completed by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. The total score can range from 0 to 54, with a higher score indicating greater severity
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 6
units on a scale | 19.0 (9.7)

5. Secondary Outcome: The Clinical Global Impression - Severity Scale
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 6
units on a scale | 4.2 (0.4)

6. Secondary Outcome: The Peabody Picture Vocabulary Test
Description: The Peabody Picture Vocabulary Test is one of the most commonly used assessment tests that measure verbal ability in standard American English vocabulary. This test has been nationally standardized using examinees from various age groups, from children to adults. Thus, the raw scores are equated to mental age, using the norms obtained from standardization. The total standard scores range from 40 (worse receptive vocabulary) to 160 (better receptive vocabulary). The scores can also be converted to percentile rank.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 6
units on a scale | 123.2 (36.6)

7. Secondary Outcome: The Social Reciprocity Scale
Description: The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows: 0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole
Number analyzed (Participants) | 6
units on a scale | 103.5 (24.4)

8. Secondary Outcome: Extra-cellular Signal-relatedness Kinase (ERK)
Description: ERK activations times, as defined as the time in minutes for ERK phosphorylation to reach the half maximal level.
Time Frame: Screen and Week 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Riluzole
Number analyzed (Participants) | 6
minutes | 2.99 (0.3)

ADVERSE EVENTS:
Time Frame: Six Weeks
Arm/Group | Riluzole
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=6)
Tiredness (General disorders) | 2 (3)
Irritability (General disorders) | 3 (3)
Worsening of Inattention (Psychiatric disorders) | 1 (1)
Appetite Reduction (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No